CLINICAL TRIAL: NCT06718660
Title: Empowering Nursing Competence in Biomedical Waste Management At El-Minia University Hospitals: a Quasi-Experimental Study
Brief Title: Empowering Nursing Competence in Biomedical Waste Management At El-Minia University Hospitals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Alaa El Din Moustafa Hamed Abd Elaleem, Lecturer of Psychiatric and mental health Nursing, Helwan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUNURSREC20241143/12
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-07

CONDITIONS: Biomedical Waste Management; Empowering Nursing Competence
Keywords: Nursing Staff; Waste management; Nursing Competence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Group (Experimental)
  Interventions: Behavioral: Tailored Educational Nursing program

INTERVENTIONS:
Behavioral: Tailored Educational Nursing program — The intervention is a structured educational program designed to enhance nursing competence in biomedical waste management at El-Minia University Hospital. It was developed based on evidence-based guidelines, national and international standards, and a detailed assessment of baseline knowledge and practices among the participating nurses.

SUMMARY:
This quasi-experimental study evaluates the impact of an educational program on improving nursing competence in biomedical waste management at El-Minia University Hospital, Egypt. The program includes three weekly sessions on waste classification, segregation, and infection control. Nurses' knowledge and practices are assessed pre- and post-intervention to measure effectiveness, aiming to enhance safe and effective waste management practices.

DETAILED DESCRIPTION:
This quasi-experimental study examines the effectiveness of an educational program designed to improve nursing competence in biomedical waste management at El-Minia University Hospital, Egypt. The program was developed following a comprehensive review of national and international guidelines, along with evidence-based literature, to address identified gaps in nurses' knowledge and practices.

The study employs a structured interview questionnaire that includes demographic details, a validated knowledge assessment tool, and a self-reported practices scale. These instruments, culturally adapted and piloted for reliability, evaluate key aspects such as understanding waste policies, segregation techniques, and adherence to infection control practices.

The intervention consists of three interactive sessions held weekly in a classroom-style setting. Sessions cover essential topics such as biomedical waste classification, associated risks, handling techniques, and infection prevention measures, with the support of illustrated educational materials.

Baseline assessments conducted during the preparatory phase guide the tailored program objectives. A follow-up evaluation one month post-intervention measures changes in participants' knowledge and practices, providing insights into the program's impact on enhancing waste management competence.

This study contributes to improving healthcare safety and compliance with biomedical waste management standards in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

Registered Nurses who have more than 6 Months of Experience and aged Between 20-60

Exclusion Criteria:

Nurses who have participated in training related to biomedical waste management within the last 12 months.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Nurses' Knowledge Regarding Biomedical Waste and Its Management | 3 months
  This outcome was assessed by using the Nurses' Knowledge Regarding Biomedical Waste and Its Management scale, which was developed by Khalil and colleagues (2024). This tool aimed to evaluate nurses' knowledge of biomedical waste and its management. It comprised 29 questions covering several key areas: knowledge of waste management policies, types of waste, hazards associated with improper waste disposal, methods of waste management, steps involved in waste handling, and locations for biomedical waste collection. Additionally, it assessed nurses' sources of information. As for the scoring system, it was as follows: two points for a fully correct answer, one point for a partially correct answer, and zero points for an incorrect or incomplete answer. Questions with only one correct answer were scored as one point for a correct response and zero for an incorrect response.

SECONDARY OUTCOMES:
Practices of Nursing Staff in Biomedical Waste Management | 3 months
  Practices of Nursing Staff in Biomedical Waste Management this was assessed by using self-reported practices of nursing staff regarding biomedical waste management, developed by Hassan and colleagues (2020) in the light of CDC guidelines. It comprised 64 items that assessed various practices, including following universal precautions when dealing with biomedical waste (10 items), adhering to color-coded segregation (9 items), following instructions on waste containers (11 items), proper disposal of sharp wastes (14 items), handling and disposing of liquid medical waste (11 items), and managing spills (9 items).

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University Hospitals, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamed AEM, Sefouhi L, Ibrahim MIT, Attia AS, Barakat AM, Elsayed EE. From knowledge to impact: revolutionizing nursing practices in biomedical waste management for sustainable healthcare excellence. BMC Nurs. 2025 Apr 29;24(1):469. doi: 10.1186/s12912-025-03073-1. PMID 40301813